CLINICAL TRIAL: NCT03311256
Title: Determination of the "Tissue Transit Time" (TTT) in the MAG3-Tc99 Diuretic Renogram for Risk Stratification of Infants With Ureteropelvic Junction Obstruction - a Multicentric Prospective Observational Study
Brief Title: Determination of the "Tissue Transit Time" (TTT)
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: TTT
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2020-11

CONDITIONS: Renal Insufficiency, Acute
Keywords: Tissue Transit Time
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tissue Transit Time — Determination of Tissue Transit Time as a prognostic and diagnostic factor

SUMMARY:
Determination of Tissue Transit Time (TTT) as a parameter with high prognostic value to predict the functional course of the differential renal function and the development of the differential renal function after pyeloplasty

DETAILED DESCRIPTION:
The ureteropelvic junction obstruction occurs in around 13% of children with antenatally diagnosed hydronephrosis. It remains a controversial topic what prognostic factors may be predictive for deterioration of the differential renal function.

The tissue transit time (TTT) in the 99mTc- MAG3 diuretic renogram seems to be a predictive factor for the deterioration of the differential renal function in these patients. We therefore analyze the tissue transit time in the 99mTc- MAG3 diuretic renogram in a prospective multicenter observational study to determine it as a prognostic and diagnostic factor. Aim of the study is to differentiate which children could be treated conservatively and which will benefit from operative pyeloplasty

ELIGIBILITY:
Inclusion Criteria:

* unilateral, isolated hydronephrosis >= grade III (SFU)
* age <= 3 months

Exclusion Criteria:

* associated malformation of the urogenital tract
* global kidney insufficiency proven by creatinine examination
* prematurity
* no informed consent

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term born infants <= 3 months of age with a unilateral, insolated hydronephrosis >= grade III (SFU)
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 3 to 6 months
  Estimation of Sensitivity and Specificity of a delayed tissue transit time as a diagnostic factor concerning worsening of the differential renal function in patients with congenital ureteropelvic junction obstruction

SECONDARY OUTCOMES:
Examination of ultrasound findings | 3 to 6 months
  Relationship between ultrasound findings and the development of the differential renal function
Examination of renal drainage | 3 to 6 months
  Relationship between initial quality of renal drainage and the development of the differential renal function
Examination of initial differential renal function | 3 to 6 months
  Relationship between initial differential renal function and the development of the differential renal function

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Luithle, MD, Principal Investigator — Universtiätsklinikum Tübingen
Locations (9):
- Germany (8):
  - Kinderchirurgische Klinik, Augsburg
  - Klinik für Kinderchirurgie und Kinderurologie, Bremen
  - Klinik für Kinderchirurgie und Kinderurologie, Dortmund
  - Kinderchirurgische Klinik, Karlsruhe
  - Zentrum für Kinder- und Jugendurologie, Mannheim
  - Klinik für Kinderchirurgie, Marburg
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinik für Kinder- und Jugendmedzin, Tübingen
- Kinderchiurgische Klinik, Luzerner Kantonsspital, Lucerne, Switzerland

REFERENCES:
- [Derived] Luithle T, Obermayr F, Dittmann H, Engel C, Etzler A, Kosch F, Menke IT, Schafer M, Schuster T, Younsi N, Fuchs J. Determination of tissue tracer transit of Technetium-99m-mercaptoacetyltriglycine diuretic renography in infants with suspected ureteropelvic junction obstruction - A multicenter prospective observational study. J Pediatr Urol. 2023 Dec;19(6):780.e1-780.e7. doi: 10.1016/j.jpurol.2023.08.029. Epub 2023 Sep 1. PMID 37718234